CLINICAL TRIAL: NCT03693391
Title: An Open-Label Study to Investigate the AMPAɣ8 Receptor Occupancy of JNJ-64140284 With the Newly Developed TARP-γ8 PET Tracer [18F]JNJ-64511070 in Healthy Men
Brief Title: A Study to Investigate Alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic Acid (AMPA Gamma 8) Receptor Occupancy of JNJ-64140284 With Newly Developed Transmembrane AMPA Receptor Regulatory Protein (TARP)-Gamma 8 Positron Emission Tomography (PET) [18F]JNJ-64511070 in Healthy Men
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: stopped because of a business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CR108508; 64140284EDI1003 (Other: Janssen Research & Development, LLC); 2018-002539-98 (EudraCT Number)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: JNJ-64140284 (Experimental): Participants in cohort 1 will receive single oral dose of JNJ-64140284 at a starting dose of 0.5 milligram (mg) under fasted conditions. The dose levels of JNJ-64140284 will be escalated sequentially based on the decisions of an independent Data Review Committee (iDRC), the clinical team and the investigator. First 3 participants will also receive an intravenous (IV) bolus injection of [18F]JNJ-64511070 at a dose of 185 megaBecquerel (MBq). Participants with no measurable brain receptor occupancy will receive second (escalated) dosing with JNJ-64140284 and subsequent positron emission tomography-computed tomography (PET-CT) scan.
  Interventions: Drug: JNJ-64140284; Drug: Fluorine-18 Labeled [18F]-JNJ-64511070
- Cohort 2: JNJ-64140284 (Experimental): Participants in cohort 2 will receive next dose level of JNJ-64140284 based upon the data-review from the previous cohort and on the decisions of an iDRC, the clinical team and the investigator. At least 3 participants will receive an IV bolus injection of [18F]JNJ-64511070 at a dose of 185 MBq. Participants with no measurable brain receptor occupancy will receive second (escalated) dosing with JNJ-64140284 and subsequent PET-CT scan.
  Interventions: Drug: JNJ-64140284; Drug: Fluorine-18 Labeled [18F]-JNJ-64511070
- Cohort 3: JNJ-64140284 (Experimental): Participants in cohort 3 will receive next dose level of JNJ-64140284 based upon the data-review from the previous cohort and on the decisions of an iDRC, the clinical team and the investigator. At least 3 participants will receive an IV bolus injection of [18F]JNJ-64511070 at a dose of 185 MBq. Participants with no measurable brain receptor occupancy will receive second (escalated) dosing with JNJ-64140284 and subsequent PET-CT scan.
  Interventions: Drug: JNJ-64140284; Drug: Fluorine-18 Labeled [18F]-JNJ-64511070
- Cohort 4: JNJ-64140284 (Experimental): Participants in cohort 4 will receive next dose level of JNJ-64140284 based upon the data-review from the previous cohort and on the decisions of an iDRC, the clinical team and the investigator. At least 3 participants will receive an IV bolus injection of [18F]JNJ-64511070 at a dose of 185 MBq. Participants with no measurable brain receptor occupancy will receive second (escalated) dosing with JNJ-64140284 and subsequent PET-CT scan.
  Interventions: Drug: JNJ-64140284; Drug: Fluorine-18 Labeled [18F]-JNJ-64511070

INTERVENTIONS:
Drug: JNJ-64140284 — Single dose of JNJ-64140284 up to 3 mg oral solution will be administered under fasted conditions.
Drug: Fluorine-18 Labeled [18F]-JNJ-64511070 — An intravenous (IV) bolus injection of 185 MegaBecquerel (MBq) [18F]JNJ-64511070 will be administered.

SUMMARY:
The purpose of this study is to measure the blocking of [18F]JNJ-64511070 binding in the brain at the time after administration of a drug when the maximum plasma concentration is reached; when the rate of absorption equals the rate of elimination (tmax) of JNJ-64140284 and determine the exposure/receptor interaction of JNJ-64140284 in healthy male participants following single oral dose administration of JNJ-64140284.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) inclusive (Body Mass Index [BMI] = weight/height^2)
* Non-smoker (not smoked for 3 months prior to screening) or/and has not used nicotine -containing products (for example, nicotine patch) for 3 months prior to screening
* Is willing to allow the investigators to place an arterial catheter in the radial artery, is assessed via physical examination (Allen Test) to be a good candidate for arterial catheter placement
* Has no history or laboratory evidence of a coagulopathy. (for participants undergoing positron emission tomography [PET] scan only)
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, in addition to the highly effective method of contraception, a man a) who is sexually active with a woman of childbearing potential and has not had vasectomy must agree to use a condom and their female partner should also use oral contraception or user independent method such as intrauterine device (IUD) or hormonal implant for at least the same duration; b) who is sexually active with a woman who is pregnant, must use a condom; c) must agree not to donate sperm

Exclusion Criteria:

* Exposed to greater than (>)1 milliSievert (mSv) of ionizing radiation participating as a participant in research studies 12 months before the start of this study
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator are acceptable
* Clinically significant abnormal physical and neurological examination, vital signs or 12-lead electrocardiogram (ECG) at screening or admission
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, liver or renal disease or obstruction to urinary flow, infection, or any other condition that the Investigator considers significant should exclude the participant. History of epilepsy or fits or unexplained black-outs
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies unless the participant has been successfully treated for HCV or HIV. Successful treatment should be confirmed by a negative ribonucleic acid (RNA) test for the virus

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Total and Regional Brain Compartmental Kinetics for Volume of Distribution (V[t]) of 18FJNJ-64511070 | Approximately up to 1 hour on Day 2
  The distribution of [18F]JNJ-64511070 in brain will be measured by positron emission tomography (PET) scans obtained along with measurement of the tracer input function with arterial samples for intact tracer and metabolites to establish the total and regional compartmental kinetics and volume of distribution (V[t]) of [18F]JNJ-64511070.
Percentage of Alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA gamma 8) Receptor Occupancy | Approximately up to 1 hour on Day 2
  Percentage of AMPAgamma8 receptor occupancy will be assessed by measuring the blocking of fluorine-18 labeled[18F]JNJ-64511070 uptake in the human brain by JNJ-64140284 using [18F]JNJ-64511070 positron emission tomography-computed tomography (PET-CT) scan and a post JNJ-64140284 scan obtained around tmax (approximately up to 1 hour on Day 2).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 6 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Change from Baseline in Electroencephalogram (EEG) Power at Day 2 | Baseline and Day 2
  EEG power spectral activity in the alpha 1, alpha 2, beta 1, beta 2, delta, theta and gamma frequency bands will be estimated for the baseline EEG recording and will be compared to the EEG power spectral activity in the same frequency bands on Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium